CLINICAL TRIAL: NCT00261924
Title: Clinical Trial to Evaluate the Therapeutic Efficacy and Safety of INTERCEPT Platelets Stored for up to Seven Days After Collection
Brief Title: Efficacy and Safety Study of Platelets Treated for Pathogen Inactivation and Stored for Up to Seven Days
Acronym: TESSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: William Reed/ Director, Clinical Research Medical Affairs, Cerus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 451-P-A-NIV
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2005-12

CONDITIONS: Thrombocytopenia
Keywords: Thrombocytopenic patients
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intercept Platelets (Experimental): Study patients receiving platelets that have been processed with the INTERCEPT pathogen inactivation system
  Interventions: Device: Transfusion of Pathogen Inactivated Platelets stored for 6-7 days
- Conventional Platelets (Active Comparator): Study patients receiving platelets processed by standard method without the INTERCEPT pathogen inactivation system
  Interventions: Device: Transfusion of Pathogen Inactivated Platelets stored for 6-7 days

INTERVENTIONS:
Device: Transfusion of Pathogen Inactivated Platelets stored for 6-7 days — pathogen inactivation of platelets for transfusion
  Other Names: INTERCEPT

SUMMARY:
Objective: To determine if platelets treated for pathogen inactivation and stored for 6 to 7 days are safe and effective compared to platelets collected by the same method, stored for the same amount of time and not treated for pathogen inactivation.

DETAILED DESCRIPTION:
Although the European Commission directive 2004/33/EC states that platelet preparations may be stored for 7 days in conjunction with detection or reduction of bacterial contamination, most blood centers store platelets for only 4 or 5 days. Extending the storage time could greatly improve platelet availability for patients while decreasing wastage of this limited resource.

ELIGIBILITY:
Inclusion Criteria:

* At least 16 years old
* Written informed consent
* Thrombocytopenia, or expected to develop thrombocytopenia requiring platelet transfusion within 15 days of randomization
* Undergoing one haematopoietic stem cell transplantation and/or admitted for treatment of acute or chronic leukaemia, lymphoma, multiple myeloma or myelodysplasia

Exclusion Criteria:

* Refractoriness to platelet transfusion
* Immune-mediated thrombocytopenia, thrombotic thrombocytopenic purpura, or hemolytic uremic syndrome
* Use of IL-11 (Neumega®) or other investigational platelet growth factor
* Disseminated intravascular coagulation (DIC)
* Clinically or radiologically detectable splenomegaly
* Previous participation in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2005-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
1 hour corrected count increment for platelets | One hour after platelet transfusion
  1-h CCI

SECONDARY OUTCOMES:
Transfusion related adverse events | 24 hours after transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Larry Corash, M.D., Study Director — Cerus Corporation
Locations (1):
- SNBTS National Science Laboratory, Edinburgh and Western General Hospital, Edinburgh, United Kingdom